CLINICAL TRIAL: NCT02962778
Title: Renin-angiotensin-system (RAS) Peptide Profiles in Patients With Treatment-resistant Arterial Hypertension (TRHT-01 Study). An Observational Single Centre Study
Brief Title: RAS Peptide Profiles in Patients With Treatment-resistant Arterial Hypertension
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: TRHT-01 Study
Record Dates: First submitted 2016-11-09; First posted 2016-11-11 (Estimated); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Hypertension
Keywords: treatment-resistant
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma samples for concentration measurement of RAS peptides and quantification of antihypertensive drug concentrations
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- treatment-resistant hypertension: patients with Treatment-resistant arterial hypertension receiving standard antihypertensive treatment with at least 3 antihypertensive agents including one diuretic

SUMMARY:
This study evaluates RAS peptides profiles in patients with treatment resistant arterial hypertension.

DETAILED DESCRIPTION:
Selective quantification of RAS peptides in human plasma triggered investigations evaluating whether RAS peptides could be used as clinical biomarkers in patients receiving antihypertensive treatment.

Drug-specific RAS profiles first characterized in healthy normotensive subjects (EKBB 255/12; ClinicalTrials.gov ID NCT01771783) are presently investigated in patients with newly diagnosed arterial hypertension (EKNZ 2015-081; clinicaltrials.gov identifier (ID) NCT02449811). With this observational study RAS peptide profiles will be characterized in patients with treatment resistant hypertension. Data generated by this study will show whether RAS peptide profiles merit further evaluation as clinical biomarkers in this complex patient group.

ELIGIBILITY:
Inclusion criteria

* Office blood pressure ≥ 140/90 mmHg and mean 24 hour blood pressure >130/80 mmHg on average, or >135/85 mmHg during the day, or > 120/70 mmHg during the night, despite concurrent use of 3 antihypertensive agents at optimal doses, including one diuretic OR
* Office blood pressure and 24 hour mean blood pressure controlled with four or more medications

  * Age ≥ 18 years
  * Ability to understand research procedures and to provide written informed consent

Exclusion criteria

* Known secondary arterial hypertension at time of inclusion or diagnosis of secondary hypertension after study inclusion during routine work-up of treatment resistant hypertension
* Known obstructive sleep apnea at time of inclusion
* History of, or clinically relevant or uncontrolled cardiovascular disease (other than arterial hypertension), namely myocardial infarction within last 3 months or valvular heart disease with clinically relevant reflux or heart failure
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the research project or compliance with the research plan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female outpatients fulfilling criteria for treatment-resistant arterial hypertension
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10-11 (Actual)

PRIMARY OUTCOMES:
RAS peptide concentrations in plasma | baseline, 4h after observed drug intake and steady-state sample

SECONDARY OUTCOMES:
Antihypertensive drug concentrations in plasma | baseline, 4h after observed drug intake and steady-state sample

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, MD, Dr., Principal Investigator — Insel Gruppe AG, University Hospital Bern
Locations (1):
- University Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
The results of this research project will be published in an appropriate scientific journal.